CLINICAL TRIAL: NCT05718557
Title: A First-in-Human, Open-label, Multicenter, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PYX-106 in Subjects With Advanced Solid Tumors
Brief Title: Study of PYX-106 in Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pyxis Oncology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PYX-106-101; 2022-002306-24 (EudraCT Number); 2023-509686-21-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor
Keywords: Solid Tumors; Advanced Solid Tumors; PYX-106; Relapsed Solid Tumors; Refractory Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PYX-106 Dose Escalation (Experimental): Participants will receive escalating doses of PYX-106 to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of PYX-106, and to determine the recommended dose(s).
  Interventions: Drug: PYX-106

INTERVENTIONS:
Drug: PYX-106 — Intravenous (IV) infusion

SUMMARY:
The primary objective of this study is to determine the recommended dose(s) of PYX-106 in participants with relapsed/refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with histologically or cytologically confirmed solid tumors who have relapsed, been non-responsive, or have developed disease progression through standard therapy.
2. Histologically or cytologically confirmed solid tumors (see details below):

   For the dose escalation, the following solid tumors are allowed in participants who have relapsed, been non-responsive, or have developed disease progression through standard therapy and in participants for whom standard of care therapy that prolongs survival is unavailable or unsuitable (according to the Investigator and after informing the Medical Monitor): non small cell lung cancer (without driver mutations/translocations), breast cancer, endometrial cancer, thyroid cancer, kidney cancer, cholangiocarcinoma, bladder cancer, colorectal cancer, and head and neck squamous cell carcinoma.
3. Clinical sites must provide archived tissue or conduct fresh tumor biopsy (formalin-fixed paraffin-embedded [FFPE]; enough to create a minimum of 14 slides). Fresh biopsy pre-treatment is preferred, archival tissue (preferably obtained within 1 year prior to the first infusion of PYX-106) is acceptable if fresh biopsy is not medically feasible, per Investigator, at Screening. Both fresh and archival tissue samples must be collected by core needle biopsy or surgical resection. Fine needle aspirates are not permitted.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
5. Participant must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 criteria (by local Investigator). Participant must have radiographic evidence of disease progression per Investigator following the most recent line of treatment.
6. Life expectancy of >3 months, in the opinion of the Investigator.

Exclusion Criteria:

1. History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; in situ cervical carcinoma, adequately treated; other adequately treated Stage 1 or 2 cancers currently in complete remission; any other cancer that has been in complete remission for >2 years or cancer of low risk of recurrence; or any treated or monitored indolent cancer that is unlikely to cause mortality in 5 years.
2. Known symptomatic brain metastases requiring >10 mg/day of prednisolone (or its equivalent) at the time of signing informed consent.
3. Continuance of toxicities due to prior anti-cancer agents that do not recover to Grade 1 prior to start of PYX-106 treatment, except for alopecia or endocrine deficiencies treated with stable hormone replacement therapy.
4. Presence of Grade ≥2 peripheral neuropathy.
5. Major surgery within 4 weeks prior to the start of PYX-106 treatment, as defined by the Investigator.
6. Received palliative radiation therapy within 14 days prior to the start of PYX-106 treatment.
7. Received a live vaccine within 28 days prior to the first dose of study treatment and while participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) | Day 1 to Day 28
Number of Participants Who Experience an Adverse Event (AE) | Day 1 up to approximately 19 months
  Type, incidence, seriousness and causality of AEs based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Any clinically significant changes in clinical laboratory parameters, vital signs, and electrocardiogram (ECG) parameters will be recorded as AEs.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of PYX-106 | Day 1 up to approximately 2 years
Time to Maximum Concentration (Tmax) of PYX-106 | Day 1 up to approximately 2 years
Area Under the Time Concentration Curve from Time 0 to the Last Quantifiable Concentration (AUC0-t) of PYX-106 | Day 1 up to approximately 2 years
Area Under the Time Concentration Curve from Time 0 to the End of the Dosing Interval (AUCtau) of PYX-106 | Day 1 up to approximately 2 years
Area Under the Time Concentration Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of PYX-106 | Day 1 up to approximately 2 years
Half Life (t1/2) of PYX-106 | Day 1 up to approximately 2 years
Objective Response Rate (ORR) | Day 1 up to approximately 2 years
Duration of Response (DOR) | Day 1 up to approximately 2 years
Progression Free Survival (PFS) | Day 1 up to approximately 2 years
Disease Control Rate (DCR) | Day 1 up to approximately 2 years
Time to Response | Day 1 up to approximately 2 years
Overall Survival (OS) | Day 1 up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (20):
- United States (11):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - SCRI- HealthOne Denver, Denver, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Lifespan - Rhode Island Hospital, Providence, Rhode Island
  - NEXT Oncology, Irving, Texas
  - NEXT Virginia, Fairfax, Virginia
- Belgium (4):
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
  - Grand Hôpital de Charleroi - Notre Dame, Charleroi, Hainaut
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
- Spain (5):
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - START Madrid - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - HM Centro Integral Oncológico Clara Campal, Madrid, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No